CLINICAL TRIAL: NCT01207063
Title: Adaptive Radiotherapy for Stage II-III Non-small Cell Lung Cancer
Brief Title: Adaptive Radiotherapy in Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRONC CONC MLD/BRONC MLD/ADA
Record Dates: First submitted 2010-07-26; First posted 2010-09-22 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Radiotherapy; NSCLC; Stage II-III non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy (Experimental)
  Interventions: Other: Radiotherapy and concurrent chemo-therapy

INTERVENTIONS:
Other: Radiotherapy and concurrent chemo-therapy — Radiotherapy and concurrent chemo-therapy

SUMMARY:
The investigators group uses an individualised radiation dose approach in which the dose is escalated up to pre-defined tissue constraints (see below). The target dose to the tumor is 69Gy. However, this dose cannot be reached in approximately 30% of the patients, even with an IMRT (Intensity Modulated Radiotherapy) technique, because the MLD (Mean Lung Dose) constraint of 20Gy is reached at a TTD (Total Treatment Dose) below 69Gy. In this study, the investigators will adapt the treatment by performing a new (PET)-CT at day 12 during radiotherapy and in case of a decreased Planning Target Volume (PTV), the dose mey be increased.

DETAILED DESCRIPTION:
Eligible patients will receive concurrent chemo-radiotherapy to the primary tumor and the initially involved mediastinal lymph nodes to an MLD (Mean Lung Dose) of 20 +/- 1Gy, irrespective of lung function.

Other dose constraints: spinal cord max: 54Gy, brachial plexus (Dmax):66Gy.

In concurrent with chemotherapy, radiotherapy will be delivered as follows:

1. First three weeks /30 fractions:twice-daily fractions of 1.5Gy, with 8h to 10h as interfraction interval, 5 days per week. Total dose: 45Gy/30 fractions.
2. Thereafter: once-daily fractions of 2.0Gy, 5 days per week until the target dose has been reached.

In sequential or radiotherapy alone schedules, twice-daily 1.8Gy with an interfraction interval of at least 8h will be delivered.

The radiation doses will be specified according to ICRU 50. Lung density corrections will be applied, as well as all standard QA procedures. Technical requirements are the same as in standard practice at MAASTRO clinic.

Chemotherapy schedules allowed:

1. 1-2 cycles induction chemotherapy: any third generation schedule is allowed. The type will be registered.
2. Concurrent part: (day 1=first day of radiotherapy)

   1. cisplatin-vinorelbine
   2. cisplatin-docetaxel
   3. cisplatin-etoposide
   4. cisplatin-pemetrexed in non-squamous histologies

Q3 week; 3 cycles

When the calculated creatinin clearance is less than 60 ml/min, cisplatin may be substituted for carboplatin.

In case the TTD(Total Treatment Dose)=69Gy cannot be reached because of a limiting MLD, a FDG-PET-CT will be performed at day 12 during radiotherapy. GTV's (Gross Tmor Volume), CTV's (Clinical Target Volume) and PTV's (Planning Target Volume) will be delineated and a new plan calculated. The endpoint will be the proportion of patients that will receive 69Gy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven NSCLC
* UICC stage I-III, or solitary metastases (<6), which are amendable for radical local treatment
* Performance status 0-2
* IMRT technique

Exclusion Criteria:

* Not NSCLC of mixed NSCLC and other histologies (e.g. small cell carcinoma)
* Stage IV, except for solitary (<6) metastases
* Performance status 3 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients able to receive 69Gy as TTD | 3 months

SECONDARY OUTCOMES:
Overall survival | 3 months
Progression free survival | 3 months
Dyspnea (CTCAE 4.0) | 3 months
Dysphagia (CTCAE 4.0) | 3 months
Patterns of recurrence | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands